CLINICAL TRIAL: NCT03501732
Title: Using Values to Enhance Inmates' Response to Substance Use and HIV Risk Feedback
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: George Mason University (Other)
Collaborators: OAR, Fairfax (Unknown); Slonky, Inc (Unknown)
Responsible Party: Principal Investigator, June Tangney, Professor, George Mason University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R34DA042974-01 (NIH)
Record Dates: First submitted 2018-03-27; First posted 2018-04-18 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Substance Use; HIV Risk Behavior
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Values Affirmation plus Risk Feedback (Experimental): Values Affirmation with Risk Feedback in substance use and HIV domains of risk
  Interventions: Behavioral: Values Affirmation; Behavioral: Risk Feedback
- Risk Feedback (Active Comparator): Sham Values Affirmation with Risk Feedback in substance use and HIV domains of risk
  Interventions: Behavioral: Risk Feedback
- Sleep Control (No Intervention): Description of sleep habits in lieu of values affirmation/sham values affirmation. No risk feedback

INTERVENTIONS:
Behavioral: Values Affirmation — Experimental Group selects two values and describes why they are important
  Arms: Values Affirmation plus Risk Feedback
Behavioral: Risk Feedback — Experimental and comparator conditions both receive normative feedback in domains of risk
  Arms: Risk Feedback; Values Affirmation plus Risk Feedback

SUMMARY:
A key component of effective offender treatment is an initial assessment of risk factors followed by feedback to facilitate problem awareness and engagement in appropriate treatment and/or behavior change. Feedback regarding areas of high risk, however, can be experienced as threatening.

The investigators propose to develop, fine-tune, and pilot-test a computerized system for risk assessment and feedback, including evaluation of a brief pre-feedback prosocial values affirmation exercise (Cohen & Sherman, 2014) aimed at decreasing defensiveness and increasing inmates' willingness to access and process risk-relevant information and to utilize post-release treatment resources, thereby reducing post-release substance misuse, HIV risk behavior, and criminal recidivism. Participants will be 170 jail inmates nearing release into the community - 20 pilot participants and 150 study participants randomly assigned to one of three conditions: (1) Values Affirmation + Personalized Risk Feedback; (2) Personalized Risk Feedback only; (3) Control. The baseline and risk assessment, values affirmation manipulation, and personalized risk feedback will be presented via touch-screen computers, requiring minimal training to administer. Analyses will assess:

1. The feasibility of utilizing a computerized system to assess and share risk information with jail inmates, including a brief values affirmation exercise to reduce defensiveness;
2. The acceptability of this approach from the perspectives of jail staff and inmates themselves;
3. The impact of the intervention on observed proximal outcomes (mechanisms of action), such as time spent viewing feedback, electing to print a copy of informational and treatment resources, and consequent changes in perceptions of risk, treatability, etc.;
4. The impact of the intervention on key post-release outcomes including engagement in relevant treatment services, substance misuse, HIV risk behaviors, re-offense and re-arrest;
5. The links between proximal outcomes (MOAs) and key post-release outcomes;
6. Potential moderators of treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient proficiency in spoken English to understand computer-assisted assessments and feedback
* post-sentencing with a sentence (i.e., less than 12 months) likely to be served out at the jail (vs. a state or federal prison) and likely to be released into the community. The invitation to participate will be timed so treatment is delivered toward the end of incarceration (within one week of release) to minimize decay of effects, and to capitalize on the motivational value of the up-coming release.

Exclusion Criteria:

* Those with detainers to other jurisdictions and to Immigration and Customs Enforcement (ICE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-08-27 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in substance use | 3 months post-release (Time 2)
  Changes in substance use -- among those who were identified at risk and who thus received feedback, pre-post incarceration changes in terms of pre-incarceration standard deviations. If more than one domain of feedback, average standard deviation change.
Changes in HIV risk behavior | 3 months post-release (Time 2)
  Changes in HIV risk behavior -- among those who were identified at risk and who thus received feedback, pre-post incarceration changes in terms of pre-incarceration standard deviations. If more than one domain of feedback (risky sex, risky needle use), average standard deviation change.

SECONDARY OUTCOMES:
Changes in accuracy of perceptions of normative risk behavior | Immediately following intervention (Time 1)
  Changes in accuracy of perceptions of normative behavior (pre-post intervention changes in terms of pre-intervention standard deviations) in areas of risk/feedback
Requests Community Resources | Immediately following intervention (Time 1)
  Choose to print a copy of community resources in domain(s) of risk
Makes Use of Community Resources | 3 months post-release (Time 2)
  Makes use of relevant community services during 3 months post-release

CONTACTS AND LOCATIONS:
Overall Officials: June P Tangney, PhD, Principal Investigator — George Mason University

IPD SHARING:
Plan to Share IPD: Yes
We will make the data and associated documentation available to researchers under a data-sharing agreement that provides for: (1) release of individually prepared datasets containing the subset of variables required to answer the requester's research question(s); (2) a commitment to using the data only for research purposes and not to attempt to identify any individual participant; (3) a commitment to securing the data using appropriate computer technology housed in a secure laboratory facility; and (4) a commitment to destroying or returning the data after analyses are completed. Because of the exceptionally sensitive nature of the data, detailed criminal history and re-arrest information and self-reports of undetected criminal behavior will not be shared. Data requests will be accepted beginning 12 months after publication of the primary findings of the proposed project.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 12 months after publication of the primary findings of the proposed project, for 5 years.
Access Criteria: Researchers who commit to using the data only for research purposes and not to attempt to identify any individual participant; who commit to securing the data using appropriate computer technology housed in a secure laboratory facility; and who commit to destroying or returning the data after analyses are completed.